CLINICAL TRIAL: NCT06541236
Title: Comparative Effectiveness of Autologous Dentin Matrix for Al-veolar Ridge Preservation
Brief Title: Alveolar Ridge Preservation After Tooth Extraction Using Autologous Dentin Matrix
Acronym: ADM for ARP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Principal Investigator, Dr. Nikolay Redko, Department of maxillo-facial and plastic sutgery, Moscow State University of Medicine and Dentistry
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Autologous Dentin Matrix (CMF)
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: To Evaluate the Quality of the Newly Formed Cortical Tissue in the Area of the Condylar Condyle Using Different Bone Grafting Materials

STUDY DESIGN:
Intervention Model Description: . The study included 80 patients in need of extraction of tooth and further dental im-plantation following proposed inclusion criteria. After selection, complex oral rehabil-itation was carried out to restore chewing function. All patients (n=80) were divided into 4 equal groups depending on the used preservative material.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of different bone grafting materials for alveolar ridge preservation of the socket (Experimental): All patients (n=80) were divided into 4 equal groups depending on the used preservative material. A total of 151 teeth were extracted. In the 1st group, the preservation was carried out using the Cerabone xenograft (Botiss, Germany). In the 2nd group, Plasma Rich in Growth Factors (PRGF) was used, obtained from the patient's venous blood 20-30 minutes before the tooth extraction (BTI Endoret, Spain). The third group consisted of patients who underwent preservation of the extracted tooth socket with crushed autologous dentin matrix (ADM) obtained from their own tooth using Smart Dentin Grinder (KometaBio Inc., USA). In the 4th group, a material based on hydroxyapatite "Kollapan-L" with lincomycin (Intermedapatit, Russia) was used as a preservation graft
  Interventions: Procedure: Alveolar Ridge Preservation After Tooth Extraction Using Autologous Dentin Matrix

INTERVENTIONS:
Procedure: Alveolar Ridge Preservation After Tooth Extraction Using Autologous Dentin Matrix — Incorporation of various bone grafting materials for alveolar ridge preservation

SUMMARY:
According to the scientific literature, the loss of any tooth can be accompanied by a pronounced resorption of the alveolar ridge in the corresponding area, which leads to the formation of various defects. In the post-extraction period, bone tissue resorption 4 months after tooth extraction is up to 45% horizontally and 43% vertically.Despite the considerable amount of research on this problem, the improvement of pre-implantation preparation of patients with adentia after tooth extraction continues to be an extremely urgent task. The solution to this problem requires a comprehensive approach based on a unified assessment of the success of dental implantation in the post-extraction zone. The aim of our study is to conduct a comprehensive comparative analysis of osteoplastic materials after preservation of the extraction wells of extracted teeth. The null hypothesis is that the ADM technique can be used in patients and the newly formed bone regenerate will be sufficient for implant placement.

DETAILED DESCRIPTION:
The study was conducted in accordance with the rules and principles of evidence-based medicine in compliance with the requirements of the Declaration of Helsinki of the World Medical Association 2013 and was approved by the Interuniversity Committee on Ethics (protocol No. 04-18 dated April 19, 2018).

The recruitment of patients and their treatment was carried out within the framework of the University Clinic of A. I. Evdokimov Moscow State University of 67 from 2018 to 2020. Study type: randomized clinical intervention prospective longitudinal study. The study included 80 patients in need of extraction of tooth and further dental implantation following proposed inclusion criteria. After selection, complex oral rehabilitation was carried out to restore chewing function. All patients (n=80) were divided into 4 equal groups depending on the used preservative material. A total of 151 teeth were extracted. In the 1st group, the preservation was carried out using the Cerabone xenograft (Botiss, Germany). In the 2nd group, Plasma Rich in Growth Factors (PRGF) was used, obtained from the patient's venous blood 20-30 minutes before the tooth extraction (BTI Endoret, Spain). The third group consisted of patients who underwent preservation of the extracted tooth socket with crushed autologous dentin matrix (ADM) obtained from their own tooth using Smart Dentin Grinder (KometaBio Inc., USA). In the 4th group, a material based on hydroxyapatite "Kollapan-L" with lincomycin (Intermedapatit, Russia) was used as a preservation graft.

4 months after tooth extraction, dental implants were installed according to the standard ITI protocol (Chen S., Buser D., 2007). In the postoperative period, a standard course of antibacterial and anti-inflammatory therapy was carried out.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, the treatment plan was discussed with each patient before surgery and an informed release form approved by the ethics committee was signed. Moreover, they met the following criteria: 1) Age from 18-70 years, 2) The presence of indications for tooth extraction: periapical periodontitis, fracture of the root or crown of the tooth without the possibility of rehabilitation, chronic periodontitis, 3) satisfactory oral hygiene.

Exclusion Criteria:

Patients under 18 years of age, pregnant women, and patients with severe comor-bidity in the stage of decompensation were not included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Level of bone persorption after Alveolar Ridge Preservation Using Autologous Dentin Matrix | 3 and 6 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Moscow State Univerciry of medicine and dentistry, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No